CLINICAL TRIAL: NCT06221670
Title: Efficacy and Safety of Toripalimab Adjuvant Therapy in High-risk Stage IA2-IB NSCLC With no Driver Alterations (EGFR or ALK) After Complete Resection: a Prospective, Single-arm Study
Brief Title: Toripalimab Therapy After Resection in High-risk Stage IA2-IB NSCLC With no Driver Alterations (EGFR or ALK)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-Toripalimab-001
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab adjuvant therapy group (Experimental): Patients must be enrolled within 8 weeks of complete surgical excision and receive Toripalimab at a dose of 240 mg intravenously (IV) once every 3 weeks for a planned duration of 1 years.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — This is a prospective, open, single-center, single-arm phase II clinical study with no driver mutations identified in the central laboratory，to evaluate the efficacy and safety of adjuvant Toripalimab therapy in completely resected stage IA2-IB non-squamous NSCLC with high-risk factors.

SUMMARY:
This is a prospective, open, single-center, single-arm phase II clinical study in non-small cell lung cancer (NSCLC) without common EGFR-sensitive mutations (Ex19del and L858R) or ALK fusion variants identified in the central laboratory. To evaluate the efficacy and safety of adjuvant Toripalimab therapy in completely resected stage IA2-IB non-squamous NSCLC with high-risk factors.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will voluntarily sign the informed consent in person, and provide the informed consent before any specific study procedures;
* Male and female, ≥18 years old;
* Primary non-squamous NSCLC confirmed histologically by the central laboratory;
* The subject was clinically confirmed as stage IA2-IB by imaging with tumor lesion size > 2 cm;
* As confirmed by the central laboratory, the tumor contains no common EGFR mutations and ALK fusion variants;
* The primary NSCLC must be completely resected by surgery, and all lesions must be removed at the end of the surgery.All surgical margins must be negative. Lobectomy can be done with open surgery or thoracoscopic (VATS);
* Central laboratory pathology confirmed solid and/or micropapillary component ≥10%, and/or STAS, and/or pleural invasion, and/or poorly differentiated, and/or complex glands ≥ 10%; PD-L1 TPS ≥ 1% in tumor tissue;
* WHO physical status score is 0~1;
* Paraffin-embedded sections (10-15 sheets), or wax blocks or fresh frozen tissue for surgical resection of the lesion should be provided;
* Adequate bone marrow reserve or organ function (demonstrated by any of the following laboratory values: absolute neutrophil count ≥1.5×10⁹/L; Platelet count ≥100×10⁹/L; Hemoglobin ≥90 g/L; Alanine aminotransferase ≤ 2.5 ULN; Aspartate aminotransferase ≤2.5 times ULN; Total bilirubin ≤ 1.5 ULN; Serum creatinine ≤1.5 ULN with creatinine clearance ≥60 mL/min [as measured or calculated by Cockcroft and Gault formulas]);
* At least 2 weeks prior to initiation of the study drug, female subjects should be using highly effective contraceptive methods, pregnancy tests must be negative, and there must be no ongoing breastfeeding prior to initiation of the drug
* Subjects voluntarily join this study, with good compliance and cooperation in safety and survival follow-up.

Exclusion Criteria:

* Exposure to other antitumor therapies before enrollment;
* Patients who only received segmental resection and wedge resection;
* Patients with any history of active autoimmune disease or autoimmune disease;
* Complicated diseases that require the use of immunosuppressive drugs; concurrent diseases that require the use of immunosuppressive agents for systemic or locally absorbable corticosteroids;
* Combined with severe heart disease, or combined with New York Heart Association (NYHA) grade 3 or 4 cardiac insufficiency;
* Any evidence of prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, or active interstitial lung disease;
* Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, any condition that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol, or active infections including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV);
* Have received preventive or attenuated vaccines within 4 weeks before the first administration;
* Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2031-03-20 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | From date of randomisation up to approximately 5 years
  DFS is defined as time from randomization to disease recurrence (determined by CT or MRI scan and/or pathologic disease on biopsy) or death (from any cause) by investigator assessment. 3-year DFS rate is Disease-Free Survival at 3 Years.

SECONDARY OUTCOMES:
DFS | From date of randomisation up to approximately 10 years
  DFS is defined as time from randomization to disease recurrence (determined by CT or MRI scan and/or pathologic disease on biopsy) or death (from any cause) by investigator assessment.
3-year OS rate | From date of randomization up to approximately 5 years
  Defined as the percentage of patients alive at 3 years, respectively, estimated from a Kaplan Meier plot of OS at the time of the primary analysis
5-year OS rate | From date of randomization up to approximately 5 years
  Defined as the percentage of patients alive at 5 years, respectively, estimated from a Kaplan Meier plot of OS at the time of the primary analysis
OS | From date of randomization up to approximately 10 years
  OS is defined as the time from the date of randomisation until death due to any cause.
Safety and tolerability in overall population | From date of randomisation up to approximately 10 years
  AEs graded by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Yue, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No